CLINICAL TRIAL: NCT05364437
Title: Pilot Clinical Trial on the Effects of Dietary Fibres on the Gut Microbiome and Metabolic Profiles in a Transgenerational Cohort
Brief Title: Investigation of the Effects of Dietary Fibres on the Gut Microbiome in a Transgenerational Cohort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 20HH5806
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Gut Health
Keywords: dietary fibres; gut microbiota; generation; metabolic profiles

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomised, cross-over
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mothers (Active Comparator): Parent to the Daughter
  Interventions: Dietary Supplement: Dietary Fibres Supplement; Dietary Supplement: Cellulose Control
- daughter (Active Comparator): Child of Mother
  Interventions: Dietary Supplement: Dietary Fibres Supplement; Dietary Supplement: Cellulose Control

INTERVENTIONS:
Dietary Supplement: Dietary Fibres Supplement — The dietary fibres supplement, which comprises of a mix of dietary fibres (inulin, pectin and oat beta-glucan) will need to be taken by participants twice daily for 2 weeks with their usual food.
Dietary Supplement: Cellulose Control — The control, which comprises of cellulose will need to be taken by participants twice daily for 2 weeks with their usual food.

SUMMARY:
Dietary fibres are complex carbohydrates present in fruit, vegetables, grains, and beans which are broken down into smaller molecules (short-chain fatty acids) in the colon by the gut microbiota. Increased intake of dietary fibres is associated with a lower risk of type 2 diabetes, obesity, or heart disease. Despite their health benefits, most people consume half of the daily recommended intake (30 grams) of dietary fibres. This trend has become more apparent in the past few decades with the advent of ultra-processed foods which are poor in dietary fibres. Since this change in dietary habits is more recent, the research team hypothesizes that older generations have a more diverse and better adapted gut microbiota at breaking down dietary fibres compared to younger generations.

The aims of this study are to examine the effects of the daily intake over four weeks of a dietary fibres supplement on the gut microbiota, metabolic profiles, and general health in a transgenerational cohort (grandmother, mother and daughter OR mother and daughter) compared to cellulose control.

DETAILED DESCRIPTION:
Eligible participants will need to take daily for 14 days a dietary fibre supplement or placebo (depending on the randomisation) followed by wash-out period of 14 days and then followed by taking daily for 14 days the opposite arm of intervention ( cellulose control or dietary fibre supplement). During the study period, participants will come to the research facility to assess the impact of these supplements on their gut microbiota, metabolic profiles and blood glucose, insulin and gut hormone levels.

ELIGIBILITY:
Inclusion Criteria:

* Any of the following groups of people (in direct descent and from the same family) Grandmother, mother and daughter Mother and daughter Grandmother and granddaughter
* Age 18-85 (inclusive)
* BMI: 18.5-30 kg/m2 (inclusive)
* Considering themselves healthy

Exclusion Criteria

* Intake of antibiotics in the past 3 months and during the study
* Intake of probiotic supplements in the past month and during the study
* Regular intake of laxatives in the past month and during the study
* Subjects with the following conditions Inflammatory Bowel Disease (IBD) Irritable Bowel Syndrome (IBS) Coeliac Disease Type 2 Diabetes Any type of cancer Autoimmune conditions Conditions that affect the liver Conditions that affect the pancreas
* Subjects who require medical intervention in the coming 3 months
* Smokers
* Shift workers
* Gluten and/or lactose intolerance
* Pregnant and lactating women
* Subjects living in care homes
* had weight changes >5% in the preceding 3 months
* Subjects who are unable to give informed consent by themselves
* Subjects who are currently participating in other clinical trials

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, PhD, RD, Principal Investigator — Imperial College London
Locations (1):
- NIHR Imperial Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Results of the study will be shared in the form of a research article or presented at scientific conferences. All results will be presented as group data rather than results for each volunteer.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers recruited by study advert Study start date 2022-10-04 Study end date 2023-04-04
Pre-assignment Details: The intervention is dietary fibres so wash out is necessary to allow the physiological measurements to return to baseline level.
Groups:
- Mothers Dietary Fibres Supplement First Then Cellulose Control: Dietary fibre mix comprising of inulin, pectin and oat beta-glucan. The mix comes in a powdered form which can be added to participants' food. Four mothers took dietary fibre mix first.
  Dietary Fibres Mix: The Fibre Mix, which comprises of a mix of dietary fibres (inulin, pectin and oat beta-glucan) will need to be taken by participants twice daily for 2 weeks with their usual food.
  This group of mothers took dietary fibre mix first and then they took the cellulose control after the wash-out period.
- Mothers Cellulose Control First Then Dietary Fibres Supplement: Control comprising of cellulose which will come in a powdered form that can be added to participants' food. Four mothers took the cellulose control first and then they took the dietary fibre mix supplement after the wash out period.
  Control: The control, which comprises of cellulose will need to be taken by participants twice daily for 2 weeks with their usual food.
- Daughters Dietary Fibres Supplement First Then Cellulose Control: Dietary fibre mix consisted of inulin, pectin and oat beta-glucan which the volunteers were able to add to their foods. The control consisted of cellulose which the participants were able to add to their foods.
  In this arm, the daughters took the dietary fibre supplement first and then they took the cellulose control following the wash-out period. Three daughters took the dietary fibre supplement first.
- Daughters Cellulose First Then Dietary Fibre Supplement.: The control consisted of cellulose which the volunteers added to their usual foods. This group of daughters took cellulose control first and then they took the dietary fibre mix after the wash-out period. In this group, five daughters took the cellulose control first.
Period: Study Period 1
Arm/Group | Mothers Dietary Fibres Supplement First Then Cellulose Control | Mothers Cellulose Control First Then Dietary Fibres Supplement | Daughters Dietary Fibres Supplement First Then Cellulose Control | Daughters Cellulose First Then Dietary Fibre Supplement.
Started | 4 | 4 | 3 | 5
Completed | 4 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout
Arm/Group | Mothers Dietary Fibres Supplement First Then Cellulose Control | Mothers Cellulose Control First Then Dietary Fibres Supplement | Daughters Dietary Fibres Supplement First Then Cellulose Control | Daughters Cellulose First Then Dietary Fibre Supplement.
Started | 4 | 4 | 3 | 5
Completed | 4 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Study Period 2
Arm/Group | Mothers Dietary Fibres Supplement First Then Cellulose Control | Mothers Cellulose Control First Then Dietary Fibres Supplement | Daughters Dietary Fibres Supplement First Then Cellulose Control | Daughters Cellulose First Then Dietary Fibre Supplement.
Started | 4 | 4 | 3 | 5
Completed | 4 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mothers: Parent to the Daughter in the placebo group
  Dietary Fibres Mix: The Fibre Mix, which comprises of a mix of dietary fibres (inulin, pectin and oat beta-glucan) will need to be taken by participants twice daily for 2 weeks with their usual food.
  Placebo: The placebo, which comprises of cellulose will need to be taken by participants twice daily for 2 weeks with their usual food.
- Daughter: Child of Mother
  Dietary Fibres Mix: The Fibre Mix, which comprises of a mix of dietary fibres (inulin, pectin and oat beta-glucan) will need to be taken by participants twice daily for 2 weeks with their usual food.
  Placebo: The placebo, which comprises of cellulose will need to be taken by participants twice daily for 2 weeks with their usual food.
- Total: Total of all reporting groups
Arm/Group | Mothers | Daughter | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  participants: <=18 years | 0 | 0 | 0
  participants: Between 18 and 65 years | 7 | 8 | 15
  participants: >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (2.1) | 26.7 (1.9) | 41.6 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 8 | 8
Fasted HbA1C [Mean (Standard Deviation); unit: mmol/l] | 37.75 (1.1) | 33.38 (0.93) | 35.56 (0.89)

OUTCOME MEASURES:

1. Primary Outcome: Stool Short-chain Fatty Acids Production Following Each Intervention Between Mothers and Daughters
Description: Changes in stool short-chain fatty acids production from baseline after each intervention (cellulose control and dietary fibre supplement) between mothers and daughters
Time Frame: 14 days
Population: Mothers and daughters data after taking the dietary fibre supplement for 14 days
Measure: Mean (Standard Error); unit: umol/g
Groups:
- Mothers Dietary Fibre Supplement: Mothers took the dietary fibre supplement for 14 days.
- Mothers Cellulose Control: Mothers took the cellulose control for 14 days.
- Daughters Dietary Fibre Supplement: Daughters took the dietary fibre supplement for 14 days
- Daughters Cellulose Control: Daughters took the cellulose control for 14 days.
Arm/Group | Mothers Dietary Fibre Supplement | Mothers Cellulose Control | Daughters Dietary Fibre Supplement | Daughters Cellulose Control
Number analyzed (Participants) | 8 | 8 | 8 | 8
umol/g | 50 (0.176) | 26 (0.709) | 41.7 (0.106) | 47.8 (0.126)

2. Secondary Outcome: Gut Microbiota Composition Changes Following Each Supplement Intake Between Mothers and Daughters
Description: Alpha diversity (a measure of the gut microbiota composition) was compared between generations after taking each dietary supplement for 14 days.
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: Urine Metabolites Comparison Between Mothers and Daughters After Taking Each Supplement
Description: Changes in urine metabolites types and levels after each generation took both supplements
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: Stool Metabolites Comparison Between Mothers and Daughters After Taking Each Supplement
Description: Changes in stool metabolites types and levels between mothers and daughters after taking each supplement. Comparisons done: mothers on dietary fibres supplement versus daughters on dietary fibre supplement and mothers on cellulose control versus daughters on cellulose control
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2025-12

5. Secondary Outcome: Blood Glucose in Mothers Compared to Daughters After Taking Each Supplement for 14 Days
Description: Fasted blood glucose levels in mothers and daughters after each generation took each supplement
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2025-12

6. Secondary Outcome: Blood Glucose for Mothers and Daughters After Taking Each Supplement for 14 Days
Description: Postprandial blood glucose levels comparison between mothers and daughters after each generation took each supplement for 14 days. The data is presented as incremental area under the curve.
Time Frame: 240 minutes
Reporting Status: Not Posted, anticipated posting 2025-12

7. Secondary Outcome: Blood Insulin Comparison Between Mothers and Daughters After Each Generation Took the Dietary Supplements
Description: Fasted blood insulin levels comparison between mothers and daughters after each generation took the dietary supplements for 14 days
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: Blood Insulin Comparison Between Mothers and Daughters After Taking Each Supplement for 14 Days
Description: Postprandial blood insulin levels comparison between mothers and daughters after each generation took the supplements (dietary fibre and cellulose) for 14 days
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2025-12

9. Secondary Outcome: Gut Hormones in Mothers Versus Daughters
Description: Fasted gut hormones levels in mothers after they took the dietary fibre supplement compared to fasted gut hormones in daughters after they took the dietary fibre supplements.
  Fasted gut hormones levels in mothers after they took the cellulose control compared to fasted gut hormones in daughters after they took the cellulose control.
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2025-12

10. Secondary Outcome: Gut Hormones in Mothers Who Took Each Dietary Supplement Versus Gut Hormones in Daughters Who Took Each Dietary Supplement
Description: Postprandial gut hormones levels were compared in mothers after they took the dietary fibre supplements against postprandial gut hormone levels in daughters after they took the dietary fibre supplement.
  Postprandial gut hormones levels were compared in mothers after they took the cellulose control against postprandial gut hormone levels in daughters after they took the cellulose control.
Time Frame: 14 days
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the time the volunteers were involved in the study. Specifically, adverse events were recorded for six weeks (two weeks on each intervention plus two weeks wash-out period).
Description: Adverse events were recorded in the study file kept in locked cabinets in the NIHR Imperial clinical research facility.
Groups:
- Dietary Fibre Supplement: Dietary fibre mix comprising of inulin, pectin and oat beta-glucan. The mix comes in a powdered form which can be added to participants' food.
  Dietary Fibres Mix: The Fibre Mix, which comprises of a mix of dietary fibres (inulin, pectin and oat beta-glucan) will need to be taken by participants twice daily for 2 weeks with their usual food.
- Cellulose Control: Control comprising of cellulose which will come in a powdered form that can be added to participants' food.
  Control: The control, which comprises of cellulose will need to be taken by participants twice daily for 2 weeks with their usual food.
Arm/Group | Dietary Fibre Supplement | Cellulose Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT05364437/Prot_SAP_000.pdf